CLINICAL TRIAL: NCT05509673
Title: Clinical Trial to Improve Wound Healing of Chronic Lower Leg Ulcers by Autologous Transplantation of Fat Tissue
Brief Title: Lipofilling for Healing of Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Collaborators: Cologne-Merheim Medical Center (CMMC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-001
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Wound Healing Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Digital analysis of wound area is masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group received a fat grafting under the wound bed and into the wound edges.
  Interventions: Other: Lipofilling (sublesional fat grafting)
- Control group (No Intervention): The control group received an injection of saline solution (0.9%) under the wound bed and into the wound edges.

INTERVENTIONS:
Other: Lipofilling (sublesional fat grafting)
  Arms: Intervention group

SUMMARY:
Chronic wounds remain a therapeutic and financial challenge for physicians and the health care systems. Innovative, cheap and effective treatment methods would be of immense value. The sublesional fat grafting could be such treatment, although the effectiveness and safety have not been assessed in large randomized clinical trials. The aim of this trial was to analyse the effect of adipose tissue on the healing of chronic lower leg wounds. For this purpose, the wounds were surgically cleaned (wound debridement) and then fat was suctioned out from the stomach or thighs and then injected into the edges of the wound and under the wounds. The wounds are covered with a foam dressing that is changed every 3-4 days. There are controls on days 3, 7, 14 and 21 after the intervention and a follow-up examination 2 months after the intervention. The primary objective is the reduction of the wound area 14 days and 2 month after intervention. Secondary objectives are pain level of the wound, bacterial colonialisation of the wound and analysis of the grafted fat tissue (ammount of mesenchymal stem cells)

ELIGIBILITY:
Inclusion Criteria:

* Patients with leg ulcers of any origin (venous, arterial, mixed arterial-venous, diabetogenic, compressive)
* Age of ulcer > 6 weeks
* Ulcer size >= 1 cm (minimum diameter)
* Ulcer / wound with complete destruction of the epidermis (including basement membrane)
* Patient age > 18 years
* Patient Consent

Exclusion Criteria:

* Pregnancy
* Exposed tendons, ligaments, or bone if maximum diameter > 2 mm
* Ulcer size > 10 cm
* Immediately preceding vacuum bandage therapy (< 2 weeks)
* Possibilities for correcting the cause of the ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-06-29 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
Reduction of wound area | 14 days and 2 month
  The reduction of the wound area from intervention to 14 days and 2 month post-intervention

SECONDARY OUTCOMES:
Pain wound | 2 month
  Subjective pain level of the patient in the area of the wound, measured by the visual analogue scale pre and post intervention
Bacterial contamination wound | 3 weeks
  Wound swabs were taken pre intervention and on days 7, 14 and 21 after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Oliver C Thamm, MD, PhD, Principal Investigator — University of Witten/Herdecke

IPD SHARING:
Plan to Share IPD: No